CLINICAL TRIAL: NCT04444479
Title: PICC Insertion With the Use of IC ECG Navigation to Confirm the PICC Tip Location Compare to Chest X-ray
Brief Title: Insertion of PICC With Intracavitary ECG Navigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PICC-07-ECG_Navigation; 07/ RVO- FNOs/ 2020 (Other Grant/Funding Number: University Hospital Ostrava); MH CZ - DRO - FNOs/2020 (Other Grant/Funding Number: Ministry of Health, Czech Republic)
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Long-term Venous Access
Keywords: peripherally inserted central catheter; ECG navigation; chest x-ray; PICC tip navigation; catheter tip location; intracavitary ECG

STUDY DESIGN:
Intervention Model Description: The study subjects enrolled in the study will be assigned to one study group. No randomization is performed.
Masking Description: No masking will be used in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PICC catheter placement (Experimental): Study subjects in whom placement of the PICC catheter is indicated
  Interventions: Other: ECG verification; Other: X-ray verification

INTERVENTIONS:
Other: ECG verification — The correct positioning of the PICC catheter tip will be verified using ECG.
Other: X-ray verification — The correct positioning of the PICC catheter tip will be verified using X-ray imaging.

SUMMARY:
The study subjects who are indicated for peripherally inserted central (PICC) catheter placement will undergo this procedure under the control of ECG, the correct position of the PICC catheter tip will be subsequently verified X-ray imaging.

DETAILED DESCRIPTION:
The study subjects who are indicated for PICC catheter placement will undergo this procedure under the control of electrocardiography (ECG), the correct position of the PICC catheter tip will be subsequently verified X-ray imaging.

Conducting this study should allow us to see the feasibility of using real-time ECG navigation, its accuracy comparing to the chest X-ray method. ´ The second goal is to eliminate chest X-ray as an obsolete method, Also the advantages and disadvantages of both methods will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* indication for establishing long-term venous access
* 18 years of age and over

Exclusion Criteria:

* oncological patients
* non-signing the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Time interval between ECG and X-ray | 2 hours
  The time elapsed between performing the ECG examination and the X-ray examination will be measured in minutes.

SECONDARY OUTCOMES:
Success-rate of correct PICC tip location | 2 hours
  The success-rate of correct PICC tip location will be determined using ECG navigation against the use of chest X-ray, and expressed as distance in centimetres from the target point.

CONTACTS AND LOCATIONS:
Overall Officials: Iveta Constantine, Bc.,MSc., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Pittiruti M, La Greca A, Scoppettuolo G. The electrocardiographic method for positioning the tip of central venous catheters. J Vasc Access. 2011 Oct-Dec;12(4):280-91. doi: 10.5301/JVA.2011.8381. PMID 21667458
- [Background] Bidgood C. Improving the patient experience with real-time PICC placement confirmation. Br J Nurs. 2016 May 26-Jun 8;25(10):539-43. doi: 10.12968/bjon.2016.25.10.539. PMID 27231736
- [Background] Johnston AJ, Holder A, Bishop SM, See TC, Streater CT. Evaluation of the Sherlock 3CG Tip Confirmation System on peripherally inserted central catheter malposition rates. Anaesthesia. 2014 Dec;69(12):1322-30. doi: 10.1111/anae.12785. Epub 2014 Jul 10. PMID 25040430